CLINICAL TRIAL: NCT04099719
Title: A GIS Mapping Exercise to Assess the Need for Injecting Equipment Provision (IEP) Services and Overdose Prevention Activities in Tayside.
Brief Title: Geographical Information System (GIS) Mapping to Assess the Need for IEP Provision in Tayside
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Sarah Donaldson, Principal Investigator, NHS Tayside
Other Study IDs: 3-010-18
Record Dates: First submitted 2019-07-04; First posted 2019-09-23 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Drug Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anyone (>16 years old) registered with services providing drug: retrospective data, no intervention to be administered

SUMMARY:
The aim of this study is to review the current provision of IEP services provided across Tayside and consider to what extent they are contributing to keeping this vulnerable population safe. The study will look at the coverage provided by the current service and map this against the known harms e.g. drugs litter finds, incidences of non-fatal overdoses and drug related deaths. This mapping process will then allow recommendations to be made in a strategic way to advise future service delivery plans to ensure that services are delivered that are reachable to the communities that need these valuable services.

DETAILED DESCRIPTION:
People who inject drugs (PWIDs) do so at significant risk to themselves due to transmission of blood borne viruses (BBV), injecting injuries, bacterial infections and drug related deaths.

NHS Tayside has a responsibility for improving the health of the population. PWIDs represent a particularly vulnerable group who experience significant health inequalities as well as stigmatisation and discriminatory attitudes.

Injecting Equipment Provision (IEP) services contribute to a reduction in BBV transmission through the provision of free sterile equipment for each injection. IEP services also provide advice on good injecting technique to avoid injecting injuries and bacterial infections. Crucially they can also provide "take home naloxone". Intramuscular injection of naloxone is a first aid emergency response for potentially fatal opiate overdoses and provides more time for emergency services to attend. Supplies of "take home naloxone" are made, along with training on overdose awareness, to those individuals at risk of opioid overdose in order to reduce the risk of fatality.

IEP services contribute to a reduction in drug related deaths by engaging with those thought to be most at risk, either through poly substance use or those who are not engaged with other services

The aim of this study is to review the current provision of IEP services provided across Tayside and consider to what extent they are contributing to keeping this vulnerable population safe. The study will look at the coverage provided by the current service and map this against the known harms e.g. drugs litter finds, incidences of non-fatal overdoses and drug related deaths. This mapping process will then allow recommendations to be made in a strategic way to advise future service delivery plans to ensure that services are delivered that are reachable to the communities that need these valuable services.

The protocol has been peer reviewed by the expert working group established to review the current provision of IEP and harm reduction and overdose awareness services across Tayside

Individual consent from patients will not be sought. The data provided by the databases will be retrospective 4 digit postcode data and will not include patient identifiable information. The data obtained will not be used in any way which may influence the care of the patient.

Data collection methods will not identify individual patients.

Researchers will be accessing information from databases which they have access to as part of their routine work. Information will remain anonymous and patient confidentiality will be upheld.

Separate consents will be sought to allow council colleagues to provide information on drug litter finds.

Anonymous 4 digit postcode data will be transferred onto Geographic Information System (GIS) maps to demonstrate coverage of services mapped against known harms (non-fatal overdoses, drug related deaths and drug litter finds). GIS maps do not identify individual postcodes.

The GIS maps will be used to identify gaps in the provision of services and provide an evidence base behind recommendations to improve service provision.

ELIGIBILITY:
Inclusion Criteria:

Anyone (>16 years old) registered with services providing drug treatment and harm reduction activities in Tayside Retrospective data from the identified databases which identifies 4 digit postcode unit of residence. All activity will be included regardless of patient characteristics.

Data will be gathered retrospectively from the past year.

Exclusion Criteria:

Data that does not identify 4 digit postcode unit of residence

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Anyone (>16 years old) registered with services providing drug treatment and harm reduction activities in Tayside
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
GIS mapping of IEP and overdose prevention activity across Tayside | 1 year
  number and 4 digit postcode location of individuals accessing IEP services, receiving Opiate Substitution Therapy from Community Pharmacy, Number and 4 digit postcode location of naloxone kits distributed, number and 4 digit postcode location of drug deaths, number and 4 digit postcode location of non fatal overdoses, number and location of drug litter finds.

SECONDARY OUTCOMES:
Construct a GIS map of the coverage of each community pharmacy in Tayside for Opiate Substitution Therapy (OST) dispensing | 1 year
  4 digit postcodes of OST prescriptions from Controlled Drug database for each community pharmacy
Construct a GIS map of the coverage of each IEP site in Tayside | 1 year
  4 digit postcodes of those accessing IEP sites recorded on NEO database
Construct a GIS map of Drug litter finds e.g. discarded needles reported to council colleagues for safe disposal | 1 year
  Postcode of locations of drug litter finds
Non-fatal overdoses mapped onto a HEAT map. | 1 year
  4 digit postcode of patients experiencing Non-fatal overdoses (NFOD) from NFOD database
Drug deaths mapped onto a HEAT map | 1 year
  4 digit postcode of those lost to Drug Deaths from Drug Death database
Take Home Naloxone supply data mapped | 1 year
  4 digit postcode information for people supplied naloxone on naloxone database

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R Donaldson, MRPharmS, Principal Investigator — NHS Tayside
Locations (1):
- Directorate of Public Health, Dundee, Tayside, United Kingdom